CLINICAL TRIAL: NCT01768325
Title: Evaluation of a New EUS-guided Needle (ProCore) Comparing to Conventional EUS-TCB Needle (Quick-Core); A Prospective Randomized, Controlled Multi-center Study.
Brief Title: Evaluation of a New EUS-guided Needle (ProCore) Comparing to EUS-TCB Needle (Quick-Core)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1104-03
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: GIST
Keywords: ProCore Needle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS-Guided biopsy needle (ProCore) (Active Comparator): Comparison of ProCore core biopsy needle to QuickCore core biopsy needle.Cook Medical core biopsy needle.
  * The number of needle passes requiring to acquire adequate specimen
  * Length of core tissue obtained
  * Diagnostic contribution of immunohistochemical staining
  * Rates of complications
  Interventions: Device: EUS-Guided biopsy needle (ProCore)
- EUS-TCB needle (Quick-Core) (Active Comparator): Comparison of core biopsy needles.
  * The number of needle passes requiring to acquire adequate specimen
  * Length of core tissue obtained
  * Diagnostic contribution of immunohistochemical staining
  * Rates of complications
  Interventions: Device: EUS-TCB needle (QuickCore) standard of care

INTERVENTIONS:
Device: EUS-TCB needle (QuickCore) standard of care — * The number of needle passes requiring to acquire adequate specimen were tallied.
  * Length of core tissue obtained
  * Diagnostic contribution of immunohistochemical staining
  * Rates of complications
  Other Names: Comparison of core biopsy needles.
  Arms: EUS-TCB needle (Quick-Core)
Device: EUS-Guided biopsy needle (ProCore) — * The number of needle passes requiring to acquire adequate specimen were tallied.
  * Length of core tissue obtained
  * Diagnostic contribution of immunohistochemical staining
  * Rates of complications
  Other Names: Comparison of core biopsy needles.
  Arms: EUS-Guided biopsy needle (ProCore)

SUMMARY:
The purpose of this study is to evaluate a new EUS-guided biopsy needle (ProCore®) comparing it to conventional EUS-TCB needle (Quick-Core®) in the diagnosis of your suspicious disorder.

This study needle (ProCore®) is a new EUS-guided biopsy needle and has been recently approved by the U.S. Food and Drug Administration (FDA) for use.

DETAILED DESCRIPTION:
Primary Objective To compare the diagnostic accuracy of new EUS histology needle (19G, ProCore, Cook Medical Inc., Winston-Salem, NC) with the conventional histology needle (19G, Quick-Core, Cook Medical Inc., Winston-Salem, NC)

Secondary Objective To compare

* The number of needle passes requiring to acquire adequate specimen
* Length of core tissue obtained
* Diagnostic contribution of immunohistochemical staining
* Rates of complications

ELIGIBILITY:
Inclusion criteria:

* Solid tumors ≥ 2 cm in size.

Exclusion criteria:

* Thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. DeWitt, M.D., Principal Investigator — Indiana University 550 N. University Hospital UH 4100 Indianapolis, IN 46202-5121
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 participants were enrolled in this study but only 78 were randomized.
Period: Overall Study
Arm/Group | Quick Core Needle | ProCore Needle
Started | 37 | 41
Completed | 37 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 78 participants competed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | QuickCore Needle | ProCore Needle | Total
Number analyzed (Participants) | 37 | 41 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 41 | 78
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 19 | 24 | 43
Region of Enrollment [Number; unit: participants]
  United States | 37 | 41 | 78

OUTCOME MEASURES:

1. Secondary Outcome: Overall Specimen Length
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Quick Core Needle: Comparison of ProCore core biopsy needle to QuickCore core biopsy needle.Cook Medical core biopsy needle
  Cook Medical core biopsy needle: Obtaining a larger specimen.
- ProCore Needle: Core biopsy needle comparison to obtain diagnostic yield.
  Cook Medical core biopsy needle: Obtaining a larger specimen.
Arm/Group | Quick Core Needle | ProCore Needle
Number analyzed (Participants) | 41 | 37
mm | 19.4 (14.1) | 4.3 (4.5)

2. Primary Outcome: Diagnostic Accuracy.
Time Frame: 36 months
Population: One patient was lost to follow up. Final diagnosis was unconfirmed.
Measure: Number; unit: Percentage of participants
Arm/Group | Quick Core Needle | ProCore Needle
Number analyzed (Participants) | 40 | 37
Percentage of participants | 88 | 62

3. Secondary Outcome: Number of Needle Passes
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: Needle passes
Arm/Group | Quick Core Needle | ProCore Needle
Number analyzed (Participants) | 41 | 37
Needle passes | 2.07 (0.72) | 2.14 (0.95)

ADVERSE EVENTS:
Time Frame: 3 years that patients were enrolled.
Arm/Group | Quick Core Needle | ProCore Needle
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/41
Other Adverse Events (participants affected / at risk) | 3/37 | 3/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quick Core Needle (N=37) | ProCore Needle (N=41)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausa/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No